CLINICAL TRIAL: NCT04256239
Title: Dignity Therapy for Terminally Ill Patients: A Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: European University of Rome (Other)
Responsible Party: Principal Investigator, Luca Iani, Associate Professor, European University of Rome
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 004/2016
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Emotional Stress; Psychological Distress; Death; Dignity
Keywords: Dignity Therapy; Terminally ill patients; Demoralization; Spiritual Well-Being; Dignity-related Distress
MeSH Terms: conditions — Stress, Psychological; Death | interventions — Dignity Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dignity Therapy Group (Experimental): Dignity Therapy is a short-term psychotherapy aimed at improving patients' sense of personhood, purpose, meaning, and self-worth and reducing psychosocial and existential distress. Therapy sessions, lasting between 20 and 60 minutes, were offered at the patients' bedside and audiotaped, and were conducted by a trained psyco-oncologist. After each therapy session, the audiotaped interview data were transcribed verbatim by a different psycho-oncologist and edited and reshaped into a written narrative by an expert in DT over the course of the next two to three days. Once the editing process was completed, another session was held to allow the therapist to read the "generativity document" to the patient and to make any editorial changes the patient deemed necessary. The final version of the generativity document was given to the patient to bequeath it to individuals of their choosing
  Interventions: Behavioral: Dignity Therapy
- Control Group (Standard Palliative Care) (No Intervention): Standard Palliative Care was performed by a multidisciplinary care team composed of a palliative doctor, a psycho-oncologist, a nurse, a physiotherapist, a healthcare assistant, a social assistant, a volunteer and a spiritual assistant, tailoring care to the needs of patients and their families.

INTERVENTIONS:
Behavioral: Dignity Therapy — Intervention aimed at enhancing patients' sense of personhood, purpose, meaning, and self-worth and reducing psychosocial and existential distress
  Arms: Dignity Therapy Group

SUMMARY:
We conducted a randomized, controlled trial of dignity therapy for terminally ill patients with the aim of reducing dignity-related distress and demoralization and improving spiritual well-being.

DETAILED DESCRIPTION:
Sample size assessment: A recent meta-analysis showed that dignity interventions reach on average effect sizes of -1.01 on emotional distress (Ho and Shin, 2014). Power analysis showed that with an alpha of 0.05 and a power of 0.80, we needed a sample of 26 participants to detect effect sizes of 1.01 and higher.

Plan for missing data: Occasional missing values were imputed by calculating, for each participant, the average score for each subscale and then replaced.

Statistical analysis plan: We conducted a 2 (group) X 3 (time [pre-treatment vs. post-treatment vs follow-up]) repeated measures multivariate analysis of variance (MANOVA) for a set of variables

ELIGIBILITY:
Inclusion Criteria:

* age over 18,
* diagnosis of life-threatening disease with a prognosis of six months or less,
* no evidence of dementia (as determined by retrospective assessments),
* the ability to read and speak Italian and provide written informed consent,
* the availability for six to seven research encounters over the period of three weeks

Exclusion Criteria:

* psychotic illness,
* dementia and severe neurological impairment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2018-02-28 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Pre-test to Post-test and Follow-up in Spiritual Well-Being, which will be reported in the outcome measure results data table as means and standard deviations. | Pre-test (before the intervention), Post-test (7-10 days after the baseline assessment), Follow-up (15-20 days after the baseline assessment).
  Spiritual well-being will be measured with the FACIT-Sp (minimum value=0; maximum value=48, with higher scores indicating a better outcome), a questionnaire assessing faith, peace and meaning

SECONDARY OUTCOMES:
Change from Pre-test to Post-test and Follow-up in Demoralization, which will be reported in the outcome measure results data table as means and standard deviations. | Pre-test (before the intervention), Post-test (7-10 days after the baseline assessment), Follow-up (15-20 days after the baseline assessment)
  Demoralization will be measured with the Demoralization Scale (minimum value=0, maximum value=32, with higher scores indicating a worse outcome), which assesses 1) Loss of Meaning and Purpose and 2) Distress and Coping Ability
Change from Pre-test to Post-test and Follow-up in Dignity-related Distress, which will be reported in the outcome measure results data table as means and standard deviations. | Pre-test (before the intervention), Post-test (7-10 days after the baseline assessment), Follow-up (15-20 days after the baseline assessment)
  Dignity-related Distress will be measured with the Patient Dignity Inventory (minimum value=25, maximum value=125, with higher scores indicating a worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Luca Iani, PhD, Principal Investigator — European University of Rome
Locations (1):
- Fondazione Sanità e Ricerca, Roma, Italy

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol
Time Frame: Data will become available after the study will be published
Access Criteria: Through the depository Figshare

REFERENCES:
- [Derived] Iani L, De Vincenzo F, Maruelli A, Chochinov HM, Ragghianti M, Durante S, Lombardo L. Dignity Therapy Helps Terminally Ill Patients Maintain a Sense of Peace: Early Results of a Randomized Controlled Trial. Front Psychol. 2020 Jun 25;11:1468. doi: 10.3389/fpsyg.2020.01468. eCollection 2020. PMID 32670169